CLINICAL TRIAL: NCT07084324
Title: Addressing Disparities: Evaluating an Executive Functioning Intervention With Spanish-speaking Neurodivergent Children and Their Families in Mexico and Colorado
Brief Title: Randomized Controlled Trial of a Spanish-language Executive Function Intervention for Neurodivergent Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-1821; 1K23MH136346-01A1 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Autism; ADHD
Keywords: executive functioning; autism; ADHD; Hispanic/Latine
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spanish Langauge Unstuck and On Target (SL-Unstuck) (Experimental): Participants in this arm will receive SL-Unstuck immediately. The intervention includes 8 weekly 90-minute clinic-based group sessions with parallel groups for children and caregivers.
  Interventions: Behavioral: Unstuck and On Target
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Unstuck and On Target — Children will receive the Unstuck and On Target (Unstuck) curriculum, a manualized cognitive-behavioral intervention that teaches executive functioning (EF) skills such as flexibility, emotional regulation, and goal-setting. Caregivers will attend concurrent Spanish-language sessions focused on understanding EF challenges and learning strategies to support their child's skills at home. Weekly home practice sheets in Spanish summarize each session and provide practical tips and activities. The program is designed to be neurodiversity-affirming and accessible to Spanish-speaking families.
  Arms: Spanish Langauge Unstuck and On Target (SL-Unstuck)

SUMMARY:
The goal of this clinical trial is to learn whether the Spanish-language version of Unstuck and On Target (SL-Unstuck), an executive functioning (EF) intervention, is feasible, acceptable, and effective for Spanish-speaking caregivers and their neurodivergent children (ages 8-11) in the U.S.. The main questions it aims to answer are:

* Is SL-Unstuck acceptable to Spanish-speaking caregivers and children?
* Does SL-Unstuck improve child EF, caregiver EF knowledge, and caregiver strain?

Researchers will compare families randomly assigned to immediate SL-Unstuck versus waitlist control to see if participating in the intervention improves EF and family outcomes.

Participants will:

* Attend 8 weekly SL-Unstuck sessions at a clinic (parallel child and caregiver groups)
* Complete pre- and post-intervention assessments on child EF, caregiver strain, and satisfaction
* Participate in a focus group to share feedback on the intervention

ELIGIBILITY:
Inclusion Criteria:

* Child is 8-11 years old.
* Child meets DSM-5 criteria for Autism Spectrum Disorder and/or ADHD
* Child has verbal skills at a 7-year-old level or greater (as measured by WASI Vocabulary and Similarities subtests)
* Caregiver endorses at least one of the following executive functioning problems:
* Difficulty accepting feedback or criticism.
* Difficulty handling frustration.
* Difficulty starting non-preferred activities.
* Frequent meltdowns.
* Not stopping a behavior after being told to stop.
* Shutting down in the face of a challenge.
* Caregiver is at least 18 years old.
* Caregiver identifies Spanish as their preferred or primary language.

Exclusion Criteria:

- Individuals will be excluded only if they do not meet one or more of the inclusion criteria listed above.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Executive Function Challenge Task | At baseline and 1 month post-implementation.
  The Executive Functioning Challenge Task deliberately tests a child's ability to utilize key executive functions like planning and flexibility by presenting scenarios that reveal potential areas of difficulty in their EF skills. The test yields Flexibility and Planning raw scores with a minimum of 0 and maximum of 8. Higher scores indicate greater impairment in executive functioning. A total executive functioning raw score is also calculated as the sum of planning and flexibility scores.
  Values below represent the change in average raw scores from baseline to post-intervention for participating children.
  Negative scores represent an overall decrease in executive functioning impairment (better outcome) while positive scores representing an increase in executive functioning impairment (worse outcome) from baseline to post when looking at the condition groups as a whole.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function Second Edition | At baseline, 1 month and 3 months post-implementation.
  The Behavior Rating Inventory of Executive Function- Second Edition is a 63-item rating scale completed by caregivers to assess executive function impairment in children. T scores have a population mean of 50 and standard deviation of 10, with a minimum score of 30 and maximum score of 95. Scales assessed included the Behavioral Regulation Index, Emotion Regulation Index and Cognitive Regulation Index, together forming an overall composite score, the Global Executive Composite. Values below represent the change in T-scores scores from baseline to post-intervention for participating children. T scores at or above 70 are considered clinically significant.
  Scores represent the change in T scores from baseline to post. Negative values represent decrease in impairment (better outcome) while positive scores representing an increase in impairment (worse outcome) from baseline to post when looking at the condition groups as a whole.
Caregiver Strain Questionnaire- Short Form 7 | At baseline and 1 month post-implementation.
  The Caregiver Strain Questionnaire-Short Form 7 is a seven item self-reported questionnaire of objective and subjective internalized caregiver strain that has been translated into Spanish. Caregivers rate how difficult or impactful different situations have been over the past month as a result of their child's behavior on a five-point Likert scale ranging from 1 "not at all" to 5 "very much." Scores are summed for a total range of 7 to 35, with higher scores indicating greater strain.
Flexibility Interference Questionnaire | At baseline and 1 month post-implementation.
  A brief questionnaire developed by researchers for parents to report how often their child's difficulties with flexibility interfere with daily adaptive functioning. It includes seven items addressing different real-world impacts, each scored on a Likert scale from 0 to 3, where 0 indicates no impact of executive function difficulties and 3 indicates severe impact. Total scores range from 0 (least interfering) to 21 (most interfering).
Executive Functions Knowledge Questionnaire | At baseline and 1 month post-implementation.
  A set of 15 true/false or multiple-choice items assesses knowledge of executive function skills and support strategies. Each question is scored as correct or incorrect, and scores are summed to yield a total number of correct responses.

IPD SHARING:
Plan to Share IPD: Yes
Deidentitifed data will be shared with NDA
Supporting Information: Study Protocol
Time Frame: Will be reported per NDA timeline
Access Criteria: Request login access to NDA